CLINICAL TRIAL: NCT05819476
Title: Boosting Open-Label Placebo Effects in Acute Induced Pain in Healthy Adults
Acronym: BOLPAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2023-00296; am23Schneider
Record Dates: First submitted 2023-03-20; First posted 2023-04-19 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Acute Pain
Keywords: Open-Label Placebo (OLP); OLP analgesia; acute pain; hyperalgesia; allodynia
MeSH Terms: conditions — Acute Pain; Hyperalgesia

STUDY DESIGN:
Intervention Model Description: The first part of this study is designed as a confirmatory, randomized, two-arm, assessor-blinded cross-over trial in a monocentric setup at the University Hospital of Basel.
  The second part is designed as a proof-of-concept, randomized, controlled, three-arm trial in a monocentric setup at the University Hospital of Basel.
Who Masked: Outcomes Assessor
Masking Description: In part 1 the assessor won't know whether subjects receive the study intervention or not (single-blinded).
  Due to organizational reasons, blinding of the assessor will not be possible in Part 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1: Visit 1 (No treatment) followed by Visit 2 (OLP intervention) (Other): In Part 1, participants will receive one injection (administration of open-label placebo injections without any active ingredient (5 ml 0.9% saline)) at twenty minutes after start of the experiment during the intervention visit 2. Visit 1 (No treatment) will be the control of the study intervention.
  Interventions: Procedure: OLP-injection; Other: Scripted Evidence-based treatment rationale; Other: Experimental model of acute pain
- Part 1: Visit 1 (OLP intervention) followed by Visit 2 (No treatment) (Other): In Part 1, participants will receive one injection (administration of open-label placebo injections without any active ingredient (5 ml 0.9% saline)) at twenty minutes after start of the experiment during the intervention visit 1. Visit 2 (No treatment) will be the control of the study intervention.
  Interventions: Procedure: OLP-injection; Other: Scripted Evidence-based treatment rationale; Other: Experimental model of acute pain
- Part 2/ Group A: 1x OLP (Control) (Other): In Part 2, the Group A (Control) receives just one single OLP injection and no repetition.
  Interventions: Procedure: OLP-injection; Other: Scripted Evidence-based treatment rationale; Other: Experimental model of acute pain
- Part 2/ Group B: 2x OLP; booster time fixed (Other): In Part 2, Group B participants will receive two injections, the first at twenty minutes after start of the experiment, and the second at a time point derived from Part 1 (if data is inconclusive; at 100 minutes).
  For every subsequent OLP administration, patients will be reminded of the inertness of the injection and that this injection might help with regulating pain.
  Interventions: Procedure: OLP-injection; Other: Scripted Evidence-based treatment rationale; Other: Experimental model of acute pain
- Part 2/ Group C: 2x OLP; booster on- demand (Other): In Part 2, Group C participants will receive two injections, the first at twenty minutes after start of the experiment, and the second on demand.
  For every subsequent OLP administration, patients will be reminded of the inertness of the injection and that this injection might help with regulating pain.
  Interventions: Procedure: OLP-injection; Other: Scripted Evidence-based treatment rationale; Other: Experimental model of acute pain

INTERVENTIONS:
Procedure: OLP-injection — Open-label placebo injections without any active ingredient (5 ml 0.9% saline). All participants will be informed that the administered injections are placebo infusions.
Other: Scripted Evidence-based treatment rationale — As a second component the intervention will consist of an evidence-based treatment rationale, which will be delivered to patients receiving the intervention prior to the OLP-injections, explaining placebo analgesia in pain in general and specifically in OLP. In the context of OLP treatments this rationale is important in order to create a mental state of positive expectations.
Other: Experimental model of acute pain — Experimental model of acute pain (simulating wound pain: this installation will apply monophasic, rectangular electrical pulses of 0.5ms duration with alternating polarity at 2 Hz frequency. The current will be increased to target a pain rating of 6 of 10 on the NRS (0 = no pain, 10 = worst imaginable pain). Three further adjustments in current will be made every 5 minutes for the next 15 minutes to compensate for habituation. This final current will be kept constant until the end of the particular experiment).

SUMMARY:
This study is to investigate the effect of open-label placebo (OLP) application on acute pain in an experimental model of acute pain (simulating wound pain: this installation will apply monophasic, rectangular electrical pulses of 0.5ms duration with alternating polarity at 2 Hz frequency. The current will be increased to target a pain rating of 6 of 10 on the NRS (0 = no pain, 10 = worst imaginable pain). Three further adjustments in current will be made every 5 minutes for the next 15 minutes to compensate for habituation. This final current will be kept constant until the end of the particular experiment).

In Part 1 duration of OLP analgesia will be examined, and onset and size of the effect will be reevaluated.

In Part 2 of this study outcomes between subjects receiving one OLP injection, subjects receiving one repetition of the injection on a fixed time point and subjects receiving one repetition of the injection on-demand will be evaluated

DETAILED DESCRIPTION:
Pain is highly prevalent in hospital settings. Standard systemic treatment for acute pain consists mainly of basic analgesia. The use of these drugs is often restricted due to their contraindications. Placebo is used nowadays to describe sham treatments and "inert" substances like sugar pills and saline injections. Placebos are proven to elicit clinically significant effects in various conditions, including pain. Ethical concerns about the use of deceptive placebos have prevented their implementation in clinical practice. A possibility to address this issue would be to prescribe placebos openly, that means, without deception. This randomized crossover study evaluates the efficacy of open-label placebo (OLP) in acute pain. Subjective pain ratings and areas of hyperalgesia and allodynia will be measured in a well-established experimental pain model (intradermal electrical stimulation model evoking pain: this installation will apply monophasic, rectangular electrical pulses of 0.5ms duration with alternating polarity at 2 Hz frequency. The current will be increased to target a pain rating of 6 of 10 on the NRS (0 = no pain, 10 = worst imaginable pain). Three further adjustments in current will be made every 5 minutes for the next 15 minutes to compensate for habituation. This final current will be kept constant until the end of the particular experiment) and analgesia elicited by OLP injections will be investigated.

In Part 1 duration of OLP analgesia will be examined, and onset and size of the effect will be reevaluated.

In Part 2 of this study outcomes between subjects receiving one OLP injection, subjects receiving one repetition of the injection on a fixed time point and subjects receiving one repetition of the injection on-demand will be evaluated (which leaves the last group a choice over when they would like to have the placebo "booster").

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (ASA Class I or II), aged 18 to 65 years
* BMI between 18 and 25kg/m2
* Able to understand the study and the NRS
* Able to give informed consent

Exclusion Criteria:

* Participation in a previous open-label placebo study; for Part 2, this includes Part 1 of this study
* Regular intake of medications or drugs potentially interfering with pain sensation (analgesics, opioids, antihistamines, calcium and potassium channel blockers, serotonin/ noradrenaline reuptake inhibitors, corticosteroids)
* Neuropathy
* Chronic pain
* Neuromuscular disease
* Dermatological disease (i.e. Atopic Dermatitis)
* Psychiatric disease
* Pregnancy / Lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Part 1: Change in Area under the Pain Curve (AUPC) | During three hours after administering an OLP
  Area under the Pain Curve (AUPC) using the numeric rating scale (NRS; 0 = no pain, 10 = worst imaginable pain) during three hours after administering an OLP
Part 2: Change in Area under the Pain Curve (AUPC) | During three hours after administering an OLP
  Area under the Pain Curve (AUPC) using the numeric rating scale (NRS; 0 = no pain, 10 = worst imaginable pain). Comparison of the AUPCs of subjects receiving just one OLP injection with subjects additionally receiving one repetition of OLP administration at a time point derived from Part 1 and subjects getting the second OLP injection on-demand.

SECONDARY OUTCOMES:
Part 1 and 2: Change in subjective pain ratings on each measurement point using the numeric rating scale (NRS) | Up to 200 minutes after electrical pain stimulation
  Change in subjective pain ratings on each measurement point using the numeric rating scale (NRS); NRS; 0 = no pain, 10 = worst imaginable pain) every five minutes after OLP administration)
Part 1 and 2: Change in Area under the Curve (AUC) of area of hyperalgesia | Up to 200 minutes after electrical pain stimulation
  Change in Area under the Curve (AUC) of area of hyperalgesia comparing the intervention and control (no treatment) visit. Pinprick hyperalgesia will be assessed every 10 minutes after OLP administration) using a 600 millinewton (mN) von Frey filament.
Part 1 and 2: Change in Area under the Curve (AUC) of area of allodynia | Up to 200 minutes after electrical pain stimulation
  Change in Area under the Curve (AUC) of area of allodynia comparing the intervention and control (no treatment) visit. Allodynia will be determined using a dry cotton swab every 10 minutes after OLP administration).

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Schneider, MD, Principal Investigator — Department of Anaesthesiology, University Hospital of Basel (USB)
Locations (1):
- University Hospital of Basel (USB); Department of Anaesthesiology, Basel, Switzerland

REFERENCES:
- [Derived] de Leeuw M, Laager M, Gaab J, Ruppen W, Schneider T. Boosting open-label placebo effects in acute induced pain in healthy adults (BOLPAP-study): study protocol of a randomized controlled trial. Front Med (Lausanne). 2024 Feb 14;11:1238878. doi: 10.3389/fmed.2024.1238878. eCollection 2024. PMID 38420356